CLINICAL TRIAL: NCT03726762
Title: Effects of Replacing Diet Beverages With Water on Type 2 Diabetic Obese Females Attending a Weight Loss Program - a Randomized, 24 Week Clinical Trial
Brief Title: Effects of Replacing Diet Beverages With Water on Weight Maintenance of Type 2 Diabetic Obese Women: 18 Months Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-307
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes; Overweight; Obese
Keywords: diet beverages; water; diabetes; weight loss; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Diabetes Mellitus; Weight Loss; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet Beverages (Experimental): 'Diet beverages' after the main meal
  Interventions: Behavioral: DBs at the end of the main meal + weight control program
- Water (Experimental): 'Water' after the main meal
  Interventions: Behavioral: Water at the end of the main meal+ weight control program

INTERVENTIONS:
Behavioral: DBs at the end of the main meal + weight control program — Subjects are asked to have 250 ml DBs at the end of their lunch as the main meal, while they are on a multidisciplinary diet plan.
  Arms: Diet Beverages
Behavioral: Water at the end of the main meal+ weight control program — Subjects are asked to have 250 ml water at the end of their lunch as the main meal, while they are on a multidisciplinary diet plan.
  Arms: Water

SUMMARY:
the present study aimed to follow up our participants in order to consider the changes in weight and anthropometric measurements after the 12-month weight maintenance as well as the total of 18 months, consisting of the previously described 24 weeks active weight loss and a further 53 weeks weight maintenance. The secondary outcome was to compare the abdominal adiposity, carbohydrate, and lipid metabolism during these periods.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic female patient with 6.5<H1AC<7.2.
* Monotherapy with Metformin.
* 18-45 years of age.
* Body mass index (BMI) between 27-35 kg/ m².
* Consume DBs regularly during their habitual diet.
* Must be able to have moderate exercise.
* Must be interested to have weight loss.

Exclusion Criteria:

* Participating in a research project involving weight loss or physical activity in the previous six months.
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medication that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Unwilling to change intake of beverages during the study period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Weight loss | 77 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose | 77 weeks
Insulin resistance (HOMA) | 77 weeks
Lipid profiles | 77 weeks
Waist circumference | 77 weeks
BMI | 77 Weeks
HA1C | 77 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hamid R Farshchi, MD, PhD, Study Chair — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ameneh Madjd, Dr, Principal Investigator — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ian A Macdonald, Prof., Principal Investigator — School of Life Sciences, The University of Nottingham; Moira A Taylor, PhD, Principal Investigator — School of Life Sciences, The University of Nottingham; Reza Malekzadeh, Prof., Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences; Alireza Delavari, MD, Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences
Locations (1):
- NovinDiet Clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided